CLINICAL TRIAL: NCT06453187
Title: Multicenter, Prospective, Randomized, Controlled Platform Trial Assessing Clinical Utility of Cellular, Acellular and Matrix-like Products (CAMPs) and Standard of Care vs SOC Alone in Hard-to-Heal Diabetic Foot and Venous Leg Ulcers.
Brief Title: A Modified Platform Trial of Multiple CAMPs for the Management of Diabetic Foot Ulcers and Venous Leg Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-WOUNDS-001
Record Dates: First submitted 2024-06-07; First posted 2024-06-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Venous Leg Ulcers with a Urinary Bladder Matrix (UBM) sheet device (Experimental): Participants will receive treatment with Urinary Bladder Matrix (UBM) sheet device, a porcine-derived extracellular matrix scaffold, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Device: Urinary Bladder Matrix (UBM) sheet device for Venous Leg Ulcers; Procedure: Standard of Care
- Diabetic Foot Ulcers with Urinary Bladder Matrix (UBM) sheet device (Experimental): Participants will receive treatment with Urinary Bladder Matrix (UBM) sheet device, a porcine-derived extracellular matrix scaffold, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Device: Urinary Bladder Matrix (UBM) sheet device for Diabetic Foot Ulcers; Procedure: Standard of Care
- Venous Leg Ulcers with AmnioExcel Plus (Experimental): Participants will receive treatment with AmnioExcel Plus, a tri-layer (amnion-chorion-amnion) dehydrated human placental membrane allograft, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Device: AmnioExcel Plus for Venous Leg Ulcers; Procedure: Standard of Care
- Diabetic Foot Ulcers with AmnioExcel Plus (Experimental): Participants will receive treatment with AmnioExcel Plus, a tri-layer (amnion-chorion-amnion) dehydrated human placental membrane allograft, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Device: AmnioExcel Plus for Diabetic Foot Ulcers; Procedure: Standard of Care
- Standard of Care (Active Comparator): Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Device: Urinary Bladder Matrix (UBM) sheet device for Venous Leg Ulcers — Application of Urinary Bladder Matrix (UBM) sheet device, a porcine-derived extracellular matrix scaffold, and participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Venous Leg Ulcers with a Urinary Bladder Matrix (UBM) sheet device
Device: Urinary Bladder Matrix (UBM) sheet device for Diabetic Foot Ulcers — Application of Urinary Bladder Matrix (UBM) sheet device, a porcine-derived extracellular matrix scaffold, and participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Diabetic Foot Ulcers with Urinary Bladder Matrix (UBM) sheet device
Device: AmnioExcel Plus for Venous Leg Ulcers — Application of AmnioExcel Plus, a tri-layer (amnion-chorion-amnion) dehydrated human placental membrane allograft, and participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Venous Leg Ulcers with AmnioExcel Plus
Device: AmnioExcel Plus for Diabetic Foot Ulcers — Application of AmnioExcel Plus, a tri-layer (amnion-chorion-amnion) dehydrated human placental membrane allograft, and participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Diabetic Foot Ulcers with AmnioExcel Plus
Procedure: Standard of Care — Participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.

SUMMARY:
The purpose of this study is to determine how well multiple CAMPs (Cellular, Acellular and Matrix-Like Products) and Standard of Care work when compared to Standard of Care alone in achieving complete closure of hard-to-heal diabetic foot and venous leg ulcers.

DETAILED DESCRIPTION:
Hard to heal Chronic wounds affect a significant percentage of patients over their lifetime. For example, diabetic foot ulcers (DFU) are a major health complication that affect up to 15% of individuals with diabetes mellitus over their lifetime. The treatment of hard to heal chronic wounds is extremely challenging as ulcers such as DFUs and Venous Leg Ulcers (VLUs) may not respond to standard of care (SC) treatment and frequently become infected.

Advanced wound products like CAMPs have become an important strategy in the treatment of hard-to-heal chronic wounds by trapping and binding the patients' own cells to rebuild the dermis layer of the skin to aid in healing.

The study will evaluate the clinical utility of Multiple CAMPs in the closure of hard to heal diabetic foot ulcers and venous leg ulcers in subjects in comparison to Standard of Care treatment.

ELIGIBILITY:
Inclusion Criteria #1: Diabetic Foot Ulcers

1. Subjects must be at least 21 years of age or older.
2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
3. At Screening Visit 1 and at Randomization, target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 20.0 cm2 measured post debridement.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care, prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the malleolus.
7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and 1.3;
   2. TBI greater or equal to 0.6;
   3. TCOM greater or equal to 40 mmHg;
   4. PVR: biphasic.
8. If the potential subject has two or more ulcers, they must be separated by at least 2 cm post debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.
10. The potential subject must consent to using the prescribed offloading method for the duration of the study.
11. The potential subject must agree to attend the weekly study visits required by the protocol.
12. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria #1: Diabetic Foot Ulcers

1. The potential subject is known to have a life expectancy of < 6 months.
2. The potential subject's target ulcer is not secondary to diabetes.
3. The target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
4. The target ulcer exposes tendon or bone.
5. There is evidence of osteomyelitis complicating the target ulcer.
6. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the Pl believes will interfere with wound healing such as biologics (monoclonal antibodies, therapeutic proteins and enzymes, gene therapies, cell therapies, cytokines and growth factors and certain vaccines) - Refer to Appendix N for a list of medications .
7. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
8. The potential subject has a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
9. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
10. Nonapplicable in this protocol version.
11. The surface area measurement of the Target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
12. The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
13. Women who are pregnant or considering becoming pregnant within the next 6 months.
14. The potential subject has end stage renal disease requiring dialysis.
15. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
16. A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
17. The target ulcer was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
18. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutrition Assessment.
19. A subject has a wound with active or latent infection as determined by the Investigator.
20. A subject with a disorder that would create unacceptable risk of post-operative complications.
21. The potential subject has a sensitivity to ethanol or porcine materials.

Inclusion Criteria #2: Venous Leg Ulcers

1. Subjects must be at least 21 years of age or older.
2. At Screening Visit 1 and at Randomization subjects must have a target ulcer with a minimum surface area of 1 cm2 and a maximum surface area of 20 cm2 measured post-debridement.
3. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
4. Nonapplicable in this protocol version.
5. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
6. If the potential subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
7. The potential subject must agree to attend the weekly study visits required by the protocol.
8. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria #2: Venous Leg Ulcers

1. The potential subject is known to have a life expectancy of < 6 months.
2. The target ulcer is infected as determined by the Investigator, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
3. The target ulcer exposes tendon or bone.
4. There is evidence of osteomyelitis complicating the target ulcer.
5. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing such as biologics (monoclonal antibodies, therapeutic proteins and enzymes, gene therapies, cell therapies, cytokines and growth factors and certain vaccines)- Refer to Appendix N for a list of medications.
6. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
7. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the Randomization visit.
8. Nonapplicable in this protocol version.
9. The surface area measurement of the target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
10. Women who are pregnant or considering becoming pregnant within the next 6 months.
11. The potential subject has end stage renal disease requiring dialysis.
12. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
13. A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
14. The potential subject was treated with hyperbaric oxygen therapy (HBOT) or CAMP in the 30 days prior to the initial screening visit.
15. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutrition Assessment
16. A subject has a wound with active or latent infection as determined by the Investigator.
17. A subject with a disorder that would create unacceptable risk of post-operative complications.
18. The potential subject has a sensitivity or allergy to ethanol or porcine materials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of complete wound closure for target ulcer | 1-12 weeks
  The percentage of target ulcers, DFU and VLU, achieving complete wound closure Complete wound closure is defined as 100% re-epithelialization of the ulcer surface without detectable exudate

SECONDARY OUTCOMES:
Time to complete wound closure for target ulcer | 1-12 weeks
  Time to closure will be determined for each treatment group and compared to SOC
Percentage of wound area reduction for target ulcer | 1-12 weeks
  Percent Area Reduction (PAR) will be calculated from measurements at Week 1 compared to measurements at week 12
Adverse Events | 1-14 weeks
  Incidence of adverse events will be evaluated weekly from the first study visit to the Closure Confirmation Visit (CCV).
Changes to pain associated with the target ulcer | 1-14 weeks
  Change in target ulcer pain assessed weekly from the first study visit to the Closure Confirmation Visit (CCV), using a 0 to 10 Pain scale with 0 = "No Pain" and 10 = "Most Intense Pain Imaginable".
Determine improvement in Quality of Life | 1-14 weeks
  Quality of Life assessed at the study randomization visit and the Closure Confirmation Visit (CCV), using a Minimal Important Difference (MID) of 0.50 based on the averaged overall score from 0 to 4 of all items the Wound Quality of Life (wQOL) checklist, with higher score indicating worse wQOL
Improvement of the Forgotten Wound Score (FWS) | 1-14 weeks
  Forgotten Wound Score (FWS) assessed at the study randomization visit and the Closure Confirmation Visit (CCV) based a 0 to 100 scale with higher indicating a high degree of "forgetting" the wound

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Serena, MD, Principal Investigator — SerenaGroup, Inc.
Locations (16):
- United States (16):
  - Phase One Clinical Trials, Inc., Bakersfield, California
  - Angel City Research, Los Angeles, California
  - Center for Clinical Research, San Francisco, California
  - ClinTrial Medical Centers, PLLC, Hamden, Connecticut
  - Alma Medical and Research Services, LLC, Hollywood, Florida
  - Symphony Research, Jacksonville, Florida
  - Lakeview Institute of Clinical Research, LLC, Leesburg, Florida
  - Denali Health Plant City, LLC, Plant City, Florida
  - Barry University Clinical Research, Tamarac, Florida
  - Denali Health, Atlanta, Georgia
  - SitePath Research, Evergreen Park, Illinois
  - Midwest Foot and Ankle Clinics, Hoffman Estates, Illinois
  - Cheyenne County Hospital, Saint Francis, Kansas
  - KUR Research, LLC, Columbia, Maryland
  - Comprehensive Wound Healing Center, Northwell Health, Lake Success, New York
  - SerenaGroup, Monroeville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No